Official Title: Examining the Effects of Stimulant Medication on Emotional Lability

in Patients with Attention Deficit Hyperactivity Disorder (ADHD)

NCT Number: NCT01415440

**Document Date:** 8/19/2019

**Study Protocol:** Youth with and without ADHD were recruited and, after the consent process, underwent diagnostic evaluations and multimodal MRI scans. Youth with ADHD were then randomized to treatment with either dexamfetamine or placebo in a 1:1 ratio. Double-bind conditions were maintained. Treatment continued for 12 weeks with dose optimized to maximize symptom improvement with minimal side effects. At the completion of treatment, youth with ADHD had a second multimodal MRI scan.

**Statistical Analysis Plan:** Image processing used the FreeSurfer platform and volumes for the amygdala and hippocampus were extracted. Treatment effects on amygdala and hippocampus volumes were tested using repeated measures factorial models. Time was a repeated measure with two levels (pre- and post-treatment), and Treatment was a between group factor with two levels (active and placebo).